CLINICAL TRIAL: NCT05846568
Title: A Phase III Clinical Trail to Evaluate the Efficacy,safety,pharmacokinetics and Immunogenicity Characteristics of GR1801 Injection for the Post-exposure Prophylaxis (PEP) of WHO Category 3 Rabies Exposure Patients.
Brief Title: Study to Evaluate GR1801's Efficacy and Safety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GR1801-003
Record Dates: First submitted 2023-04-06; First posted 2023-05-06 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2023-09

CONDITIONS: Rabies Post-exposure Prophylaxis
Keywords: Rabies; Rabies virus neutralizing antibodies; Post-exposure prophylaxis
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Intervention Model Description: 1200 patients aged 18 and above with WHO Category III rabies exposure should be enrolled as planned and randomly assigned to the GR1801 injection group and the HRIG group based on a ratio of 3: 1. The random stratification factors include time of exposure (within or beyond 24 hours), bite location (above or below the neck), and number of bites (1 or more).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group: GR1801+Rabies vaccine(CHENGDA PHARMACEUTICALS) (Experimental): GR1801 injections are administered by wound infiltration injection or by intramuscular injection.GR1801 injections are a bispecific monoclonal antibody that exhibit a wide spectrum of activity against various wild-type rabies strains in vitro.
  Dosage form:2mg/1mL/vial, liquid, Dosage: 0.05mg/kg of GR1801 Frequency/duration: at Day 0.
  Rabies vaccine should be administered in deltoid muscle Dosage form: >=2.5 IU, freeze-dried vaccine, 0.5 mL after reconstitution, Frequency/duration: at Day 0, 3, 7, 14, 28.
  Interventions: Biological: GR1801; Biological: Rabies Vaccine
- Control Group:HRIG（BOYA-BIO）+Rabies vaccine(CHENGDA PHARMACEUTICALS) (Active Comparator): HRIG is administered by wound infiltration injection or by intramuscular injection. Dosage form: 200 IU/2mL/vial, liquid, Dosage: 20 IU/kg, Frequency/duration: at Day 0.
  Rabies vaccine should be administered in deltoid muscle Dosage form: >=2.5 IU, freeze-dried vaccine, 0.5 mL after reconstitution, Frequency/duration: at Day 0, 3, 7, 14, 28.
  Interventions: Biological: Human Rabies Immunoglobulin(HRIG); Biological: Rabies Vaccine

INTERVENTIONS:
Biological: GR1801 — The injection solution GR1801 does not contain preservatives. The excipients include histidine/histidine hydrochloride (20mM), trehalose (90 mg/mL), disodium EDTA (0.372mg/mL) and polysorbate 80 (0.5 mg/mL). The pH value is 5.8 and each bottle contains 2mg of GR1801 protein. The packaging material is a borosilicate glass tube injection bottle (2mL) with a halogenated butyl rubber stopper for injection and an aluminum-plastic composite cap for antibiotic bottles.
  Arms: Experimental Group: GR1801+Rabies vaccine(CHENGDA PHARMACEUTICALS)
Biological: Human Rabies Immunoglobulin(HRIG) — The HRIG is a Chinese licensed Human Rabies Immunoglobulin produced by BOYA-BIO, which are derived from human plasma, and then purified and filled in the injectable vial form.
  Arms: Control Group:HRIG（BOYA-BIO）+Rabies vaccine(CHENGDA PHARMACEUTICALS)
Biological: Rabies Vaccine — The Chinese licensed freeze-dried rabies vaccine produced by CHENGDA PHARMACEUTICALS for human use (Vero Cells) which is indicated for the rabies Post-exposure Prophylaxis (PEP) .

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of GR1801 injection with Human Rabies Immunoglobulin(HRIG) in patients with WHO Category 3 rabies exposure.

Patients will receive GR1801 injection or HRIG. Each group will receive rabies vaccine as the WHO Essen regime after Study Drug.

DETAILED DESCRIPTION:
This is a randomized, double-blind, Human Rabies Immunoglobulin(HRIG) controlled Phase III clinical trial evaluating the efficacy, safety, pharmacokinetic and immunogenicity of GR1801 injection as a part of post-exposure prophylaxis (PEP) in patients with WHO Category 3 rabies exposure who have met all inclusion/exclusion criteria for their treatment group.

1200 patients aged 18 and above with WHO Category III rabies exposure should be enrolled as planned and randomly assigned to the experimental group and the control group based on a ratio of 3: 1. The random stratification factors include time of exposure (within or beyond 24 hours), bite location (above or below the neck), and number of bites (1 or more).

All the patients should receive wound infiltration injection of GR1801 or HRIG on Study Day 0 (wound conditions should be described and recorded both before and post injection by photos, including diameter, depth, expansion treatment, etc.), and should also receive intramuscular injection of one dose of the freeze-dried rabies vaccine for human use (Vero cells) into the deltoid muscle after the infiltration injection. Patients should also be given one dose of the freeze-dried rabies vaccine for human use (Vero cells) on Study Days 3, 7, 14, and 28 respectively according to the WHO Essen regime.

Rabies virus neutralizing antibodies (RVNA) should be collected 9 times from each subject prior to administration and on Study Day1, 3, 5, 7, 14, 42, 90, 365 post administration of Study Drug. RVNA should be assayed through rapid fluorescence focus inhibition test (RFFIT). The occurrence of rabies and survival conditions should be collected through every follow-up visit.

Adverse events should be classified in accordance with solicited adverse events and unsolicited adverse events. Solicited adverse events include local adverse events (such as injection sites pain, induration, swelling, redness, rash and pruritus) and systemic adverse events (such as fever, hypersensitivity, headache, fatigue, nausea, vomiting, arthralgia and myalgia). Unsolicited adverse events are those except solicited adverse events or solicited adverse events beyond 7 days after the first administration.

Solicited adverse events should be collected 7 days after the first administration. Unsolicited adverse events should be collected in 3 months after the first administration and serious adverse events(SAE) should be collected throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese males or females aged 18 years or above on Study Day 0 with legal identification documents and plan to live in the local area during the study;
2. WHO Category III rabies exposure；
3. Those who have an armpit temperature ≤ 37.0 °C；
4. Completed written informed consent process, signed the informed consent forms and Agreed to complete all follow-ups.

Exclusion Criteria:

1. WHO Category III rabies exposure but received wound suture treatment;
2. WHO Category III rabies exposure over 72 hours;
3. Previous receipt of rabies vaccination or rabies passive immunization;
4. History of bitten by animals such as dogs, cats, bats etc. within the 6 months before the Study Day 0;
5. History of any severe allergy for vaccination;
6. Had fever (armpit temperature ≥ 38.5 °C) or received any antipyretic, analgesic or anti-allergic drug within 3 days before Study Day 0;
7. History of severe autoimmune diseases;
8. History of any severe neurological disease；
9. History of receiving any immunoglobulin or vaccine within 30 days before Study Day 0, or plan to use any such product during the study;
10. History of addiction to any narcotic, alcohol or drugs;
11. Previous receipt of any study product (drug, vaccine, biological product or device) within 6 months before Study Day 0, or plan to participate in any other clinical study during this study period;
12. Females who are pregnant or with urine pregnancy test positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the Geometric mean RVNA Concentration (accessd by Rapid Fluorescent Foci Inhibition Test(RIFFIT)) for GR1801 recipients is non-inferior to the Geometric mean RVNA Concentration for HRIG recipients on Study Day 7. | 7 days
  RVNA（Rabies Virus Neutralizing Antibodies） geometric mean concentration of GR1801 recipients and HRIG recipients in combination with rabies vaccines.
To evaluate the percentage of subjects with RVNA concentration ≥ 0.5 IU/mL on Study Day 14 in GR1801 recipients is non-inferior to the percentage of subjects with RVNA concentration ≥ 0.5 IU/mL for HRIG. | 14 days
  The percentage of subjects with the RVNA geometric mean concentration ≥ 0.5 IU/mL in GR1801 recipients and HRIG recipients in combination with rabies vaccines.
To evaluate the rabies post-exposure protection rate for GR1801 recipients is non-inferior to the protection rate for HRIG recipients on Study Day 365. | 365 days
  The percentage of subjects with no case of rabies death in GR1801 recipients and HRIG recipients in combination with rabies vaccines.

SECONDARY OUTCOMES:
To evaluate the rabies post-exposure morbidity of GR1801 compared to HRIG within 90 days and 365 days after administration. | 365 days
  The percentage of subjects with probable or confirmed cases of rabies.
To evaluate the rabies post-exposure mortality of GR1801 compared to HRIG within 90 days and 365 days after administration. | 365 days
  The percentage of subjects with cases of rabies death.
To evaluate the rabies post-exposure survival rate of GR1801 compared to HRIG within 90 days and 365 days after administration. | 365 days
  The percentage of subjects with rabies-free survival.
To evaluate the Geometric mean RVNA Concentration of GR1801 compared to HRIG within 1,3,5,14,42,90 and 365 days after administration. | 365 days
  RVNA geometric mean concentration.
To evaluate the percentage of subjects with RVNA concentration ≥ 0.5 IU/mL of GR1801 compared to HRIG within 1,3,5,7,42,90 and 365 days after administration. | 365 days
  The percentage of subjects with RVNA geometric mean concentration ≥ 0.5 IU/mL.
To evaluate the detection rate of RVNA concentration of GR1801 compared to HRIG within 1,3,5,7,14,42,90 and 365 days after administration. | 365 days
  The percentage of subjects whose RVNA geometric mean concentration are below the quantization limit.
To evaluate the safety of GR1801 compared to HRIG within 365 days. | 365 days
  Number of participants with treatment-related adverse events or serious adverse events as assessed by CTCAE v5.0
To evaluate the peak plasma concentration(Cmax) of GR1801 within 365 days. | 365 days
  The peak plasma concentration of GR1801 will be estimated at D3,D7,D14 and D42,using non compartmental analysis.
To evaluate the Area under the plasma concentration versus time curve (AUC0-last,AUC0-inf) of GR1801 within 365 days. | 365 days
  The Area under the plasma concentration versus time curve (AUC0-last,AUC0-inf) of GR1801 will be estimated at D3,D7,D14 and D42,using non compartmental analysis.
To evaluate the immunogenicity of GR1801 within 365 days. | 365 days
  To assess the anti-drug-antibodies (ADA) and neutralizing antibodies (NAb) of GR1801.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqiang Liu, PHD, Principal Investigator — Yunnan Province Center for Disease Control and Prevention (CDC)
Locations (1):
- Center for Disease Control and Prevention (CDC), Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No